CLINICAL TRIAL: NCT02788825
Title: STHLM3-MR: Comparing Standard With Targeted Prostate Biopsies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Tobias Nordström, MD PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STHLM3MR-1
Record Dates: First submitted 2016-05-11; First posted 2016-06-02 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Targeted biopsies using Magnetic Resonance Imaging guiding — Prostate biopsies targeted by findings on MRI where findings are classified according to PI-RADS v2.

SUMMARY:
Prostate cancer is a leading cause of cancer death among men in the Western world. Early detection of prostate cancer has been shown to decrease mortality, but has limitations with low specificity leading to unnecessary biopsies and over-diagnosis of low-risk cancers. The STHLM3 trial has paved the way for improved specificity in early detection of prostate cancer using the blood-based STHLM3 test for identifying men at increased risk of harbouring significant prostate cancer.

Targeted prostate biopsies based on MRI images have been shown to increase sensitivity of high-grade cancers compared to the currently used systematic biopsies, but existing evidence are contradictory and not free from methodological flaws.

The primary aim of STHLM3-MR/Fusion is to increase the specificity in early detection of prostate cancer without decreasing the sensitivity of aggressive prostate cancers by introducing targeted prostate biopsies and comparing to traditional prostate biopsies. The primary endpoints are the number of performed biopsies and the number of detected high-grade prostate cancers defined as Gleason 7 or higher. Secondary endpoints include the number of low risk prostate cancers diagnosed and the proportion of patients with up-or downgraded disease after assessment of prostatectomy specimen. Additional aims include to assess the health economic consequences of implementing MRI based prostate cancer diagnostics and to improve the quality and effectiveness of prostate cancer diagnosis in the routine health care in Stockholm.

The STHLM3-MR/Fusion project will be performed in two separate phases, analyzed separately. Based on power calculations, approximately 500 planned for prostate biopsies will be included in the first phase. Men who have previously been diagnosed with prostate cancer may not take part in the study. The study period of Phase 1 is March 2016 to January 2017. The second phase will start in autumn 2016 and end by December 2017.

ELIGIBILITY:
Inclusion Criteria:

* Men age 45-75 years referred to any of the participating urological centers for prostate biopsies

Exclusion Criteria:

* A prior diagnosis of prostate cancer (ICD-9 C61)
* Severe illnesses such as metastatic cancers, severe cardio-vascular disease or dementia
* Contraindications for magnetic resonance imaging (MRI) eg pacemaker, magnetic cerebral clips, cochlear implants or severe claustrophobia.

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 687 (Actual)
Dates: Start 2016-04; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Estimated number of targeted biopsies needed to maintain Gleason sum 7 sensitivity as compared with systematic biopsies. | Assessed after 500 (paired) biopsies are performed in Stockholm. Timeframe: from April 2016 to April 2017, up to 1 year
Total number Gleason sum ≥7 tumours detected by targeted and systematic biopsies, respectively | Assessed after 500 (paired) biopsies are performed in Stockholm. Timeframe: from April 2016 to April 2017, up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Nordström, MD PhD, Principal Investigator — Dpt Medical Epidemiology and Biostatistics, Karolinska Institutet
Locations (2):
- Aleris Oslo, Oslo, Norway
- Karolinska Universitetssjukhuset, Solna, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lantz A, Haug ES, Picker W, Crippa A, Jaderling F, Mortezavi A, Nordstrom T. Effect of information on prostate biopsy history on biopsy outcomes in the era of MRI-targeted biopsies. World J Urol. 2021 Apr;39(4):1153-1159. doi: 10.1007/s00345-020-03277-x. Epub 2020 May 29. PMID 32472278
- See also: Website STHLM3 projects — http://sthlm3.se